CLINICAL TRIAL: NCT03516734
Title: The Effect of Iron-fortified Lentils on the Iron (Fe) Status Among the Adolescent Girls in Bangladesh- a Double-blind Randomized Controlled Trial
Brief Title: Iron-fortified Lentils to Improve Iron (Fe) Status in Bangladesh
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Carol Henry (Other)
Collaborators: Brac (Other); Marywood University (Other); Nutrition International (Other)
Responsible Party: Sponsor-Investigator, Carol Henry, Professor, University of Saskatchewan
Organization: University of Saskatchewan (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: Bio# 17-177
Record Dates: First submitted 2018-02-28; First posted 2018-05-04 (Actual); Last update posted 2020-11-04 (Actual); Status verified 2020-11

CONDITIONS: Anemia, Iron-Deficiency; Cognitive Performance; Iron-deficiency
Keywords: Iron deficiency; Food-based dietary intervention
MeSH Terms: conditions — Anemia, Iron-Deficiency; Iron Deficiencies

STUDY DESIGN:
Intervention Model Description: Thick preparation of cooked Iron-fortified lentils (37.5gm raw lentil) will be provided. There will be three lentils based dietary intervention arm in this efficacy trial. Arm 1 will be intervened with iron-fortified lentils, Arm 2 will be non-iron fortified lentils, and Arm 3 arm will be the usual intake of lentil (no additional lentil). Arm 2 will be served as a comparison group and arm 3 will be served as control group.
Who Masked: Participant, Care Provider, Investigator
Masking Description: Participants, care provider, and investigators will be masked on the distribution of iron-fortified lentil among 3 different adolescent group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Iron fortified lentils (Experimental): Lentils will be fortified with iron in the lab setting at the Crop Development Center (CDC) of The University of Saskatchewan, Canada. The study will fortify lentil by spraying iron fortificant NaFeEDTA solution. A small sprayer will be placed at the beginning of the lentil polishing machine at a commercial lentil mill located near Saskatoon, Canada. The iron solution will be applied as a fine mist which will be absorbed into the lentil as it travels through the polishing drum. As the fortified lentil leaves the drum it will be bagged in 20 kg food grade bags. The expected concentration of Fe in the final product will be approximately 21 mg/100 g of lentil (fortified with NaFeEDTA solution with 1600 ppm of Fe).
  Interventions: Dietary Supplement: Iron fortified lentils
- Non iron-fortified lentils (Active Comparator): It will be the same Saskatchewan (province of Canada) grown small cotyledon color lentil (Iron content 75-90ppm) without the iron fortification.
  Interventions: Other: Non Iron-fortified lentils
- Usual Intake (no intervention) (Placebo Comparator): It will be the usual intake of lentil- no additional lentil will be provided. However, participants will be free to consume lentils from anywhere (homemade or restaurants) if they want to, except our fortified lentils.
  Interventions: Other: Usual Intake

INTERVENTIONS:
Dietary Supplement: Iron fortified lentils — Lentils will be iron-fortified using NaFeEDTA iron fortificants
  Arms: Iron fortified lentils
Other: Non Iron-fortified lentils — Non-fortified lentils will be provided
  Arms: Non iron-fortified lentils
Other: Usual Intake — No lentils will be provided.
  Arms: Usual Intake (no intervention)

SUMMARY:
We designed a double-blind, community-based, cluster-randomized control trial which will test to establish novel evidence on the efficacy of iron-fortified lentil in improving body Fe status of non-pregnant adolescents in rural Mymensingh district of Bangladesh. Lentils will be fortified with iron in the lab setting at the Crop Development Center (CDC) of the University of Saskatchewan in Canada. There will be three lentils based dietary intervention arm in this efficacy trial. Arm 1 will be intervened with iron-fortified lentils, Arm 2 will be non-iron fortified lentils, and Arm 3 arm will be the usual intake of lentil (no additional lentil). Arm 2 will be served as a comparison group and arm 3 will be served as control group. A total of 420 adolescent girls (including 20% drop-outs) - aged 10 - 17y; non-smoking, not pregnant, not breastfeeding, and generally healthy will be included in each arm - a total of 1260 adolescent girls in all three arms. Participating adolescents will be served thick preparation of cooked lentils (37.5gm raw lentil) 5 days a week for 85 feeding days (around 4+months). Socio-demographic characteristics, household food security status, and adolescent food habits will be collected at baseline and endline data point. Furthermore, venous blood will be collected to measure adolescents' Fe status at baseline, midline, and endline for 85 feeding days (5 days a week)- approx. 4+ months. In addition, Ravens Progressive Matrices will be used for non-verbal measurement of the cognitive ability of advanced observation and thinking skills specific to capacity for analyzing and solving problems, abstract reasoning, and the ability to learn of the adolescents. Both descriptive and inferential statistics will be used for this study. Serum ferritin level and cognitive performance is the primary outcome. The trial expects that the supplemental Fe from the iron-fortified lentils will improve body Fe status and cognitive performance after controlling for baseline Fe status and dietary Fe intake in this group of adolescent girls. The secondary outcome is the participants' anthropometries. Considering the amount of plant protein from lentils that need to be consumed to for the study, it is expected to have significant improvement in growth of the participants which will lead to increased productivity.

DETAILED DESCRIPTION:
The study will be implemented in collaboration with BRAC (Bangladesh Rural Advancement Committee) is one of the top-ranked most effective multinational non-government organization (NGO) in the world- headquarter based in Dhaka, Bangladesh. Among many development programmes, BRAC has a specific programme for adolescents- named 'BRAC Adolescent Development Programme' which formed adolescent clubs as a part of their project. These clubs targeted all adolescent girls in the community regardless of their school attendance, marital status, pregnancy, or socio-economic status. The clubs provide a unique place and opportunity for adolescents to socialize both in rural and urban settings. Each club comprises of 25-40 adolescents, mainly girls and a few boys member between ages 10 to 19 years. These clubs operate in afternoons in BRAC schools, while in the absence of such facilities, a room is rented locally by BRAC.The efficacy study will be conducted at the BRAC's Adolescent Clubs. The adolescent Clubs will be selected from 4 Upazilas i.e., Muktagacha, Nanadail or Mymensingh Sadar (Central), Bhaluka, Gaffargaon of Mymensingh district in Bangladesh. There will be three lentils based dietary intervention arm in this efficacy trial. Arm 1 will be intervened with iron-fortified lentils, the 2nd arm will be non-iron fortified lentils, and 3rd arm will be the usual intake of lentil (no additional lentil). Arm 2 will be served as a comparison group and arm 3 will be served as control group. Considering the lower estimation on the expected difference in mean serum ferritin (5mgm/L) with 80% power at 0.05 significance level, Intra Cluster Correlation (ICC) 0.025, a total of 59 cluster will be selected (each club will be treated as a cluster) where a total of 11 eligible adolescent girls will be selected from each cluster. A total of 335 adolescent girls will be placed in each of the intervention arms. The sample size was further incremented to minimize 20% lost to follow-up (resulting 420 in total) during the intervention period of 85 feeding days (approx. 4 months). Thus, the total sample size would be 1252 adolescent girls. A total of 20 adolescent clubs (420 adolescent girls - including 20% drop-outs) will be included in each arm - a total of 1252 adolescent girls in three arms. Participating adolescents will be served thick preparation of cooked lentils (37.5gm raw lentil) 5 days a week for 85 feeding days (around 4+months). In a typical week, the BRAC adolescent club run for 2 days a week (Thursday and any other day). As this study proposes to serve daal 5 days a week, the research team will invite participants to visit the clubs for extra 3 days and consume the cooked lentil/daal. BRAC field level staff will encourage adolescent girls to come to clubs and also their parent to allow them to join the club for consuming dal. These adolescent girls reside in the area near the clubs. The researchers, therefore, assume that there will be full participation in non-club days.

All adolescent girls will be enrolled in the study, will be tested for parasites and be de-wormed prior data collection. Baseline, midpoint and endpoint data collection will include venous blood samples to measure Fe status, anthropometry, and cognitive outcomes. Each of the survey (baseline and endline) survey would take around 30 min per participants. However, in the midline, only venous blood samples will be collected to measure body iron status. Fe status measurement will include hemoglobin, hematocrit (volume of red blood cells), serum ferritin, soluble transferrin receptor (sTfR), C-reactive protein and imputed total body Fe (Aim 1). Height, weight, mid-upper arm circumference (MUAC), and total serum ferritin (TSF) of adolescents will be measured regularly (Baseline and endline) during the study to determine the change in growth. Ravens Progressive Matrices (RPM) and Cambridge Neuropsychological Test Automated Battery (CANTAB) assessments will be used for non-verbal measurement of the cognitive ability of advanced observation and thinking skills specific to capacity for analyzing and solving problems, abstract reasoning, and the ability to learn. Two rounds of data collection in the baseline and endline will include information on socio-demographic characteristics, household food security status, and adolescent food habits (FFQ). Periodic data collection will be carried out in order to track the smooth intervention with defined intervals (every month) on the compliance of the respondents, participants' morbidity including parasitic infestation, menstruation, fortified lentil distribution efficiency, fortified lentil stock, and other explanatory variables. Process evaluation of intervention performance will be conducted in a selected number of adolescent clubs to understand if the interventions are implemented as planned. The process evaluation will provide information related to intervention impact pathway and immediate feedback to the project implementers. In addition, it will help to interpret the research findings. A venous blood sample (approx. 10ml) will then be collected by a well-trained phlebotomist from each of the participants using lithium heparinized vacutainer following aseptic procedure and using disposable syringe and needle. Vacutainers will be carried to the nearest field laboratory in an ice box for serum separation and which will then be stored at 2-8 degree Celsius (°C). All plasma samples will be shipped to central laboratory of International Centre for Diarrhoeal Disease Research, Bangladesh (ICDDR,B) based in Dhaka within 72 hours of collection where the samples will be analyzed. The blood collection per participants will take around 10 min.

ELIGIBILITY:
Inclusion Criteria:

* Adolescent girls who attend the BRAC adolescent clubs
* Age between 10 -17 years
* Non-smoking
* Not pregnant
* Not breastfeeding
* Generally healthy.

Exclusion Criteria:

* Unwilling to participate
* Active illness during recruitment
* Known case of Infectious disease

Ages: 10 Years to 17 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child
Gender Based: Yes — Participant eligibility is based on self-representation of gender identity.
Enrollment: 1252 (Estimated)
Dates: Start 2018-09-30 (Actual); Primary Completion 2019-04-09 (Actual); Study Completion 2021-04-30 (Estimated)

PRIMARY OUTCOMES:
Changes in Serum ferritin level (micrograms per liter) | 85 feeding days
  Body Fe status (micrograms per liter) will be measured at baseline, midline, and endline at 85 feeding days (5 days a week)- approx. 4+ months

SECONDARY OUTCOMES:
Cognitive performance [(non-verbal measurement), # items correct out of 60-item test] | 85 feeding days (change from baseline cognitive ability at endpoint)
  Standard Progressive Matrices will be used for non-verbal measurement of the cognitive ability of advanced observation and thinking skills specific to capacity for analyzing and solving problems, abstract reasoning, and the ability to learn. The booklet comprises five sets (A to E) of 12 items each (e.g., A1 through A12), with items within a set becoming increasingly difficult, requiring ever greater cognitive capacity to encode and analyze information. All items are presented in black ink on a white background.
  Higher the number of correct answers higher the cognitive ability.
  It would take around 45 minutes per participant.
Attention assessment (# of correct response) | 85 feeding days (change from baseline attention at endpoint)
  Attention assessment (# of correct response) test will be administered via The Cambridge Neuropsychological Test Automated Battery (CANTAB) [www.cambridgecognition.com].
  Higher number of correct responses would be treated as better performer.
  Tests would take around 45 minutes per adolescent.
Visual memory assessment [Time (seconds and milliseconds)] | 85 feeding days (change from baseline visual memory at endpoint)
  Visual memory assessment by test administered via The Cambridge Neuropsychological Test Automated Battery (CANTAB) (www.cambridgecognition.com).
  Correct responses within the shorter time would be treated as better performer.
  Tests would take around 45 minutes per adolescent.
Height (centimetre) | 85 feeding days
  Adolescents height will be measured in centimetre (cm).
Body weight (kilogram) | 85 feeding days
  Adolescents weight will be measured in kilogram (kg)
Waist Circumference (centimetre) | 85 feeding days
  Adolescents waist circumference will be measured in centimetre (cm).
Mid-upper arm circumference (centimetre) | 85 feeding days
  Adolescents mid-upper arm circumference will be measured in centimetre (cm).
Hip circumference (centimetre) | 85 feeding days
  Adolescents hip circumference will be measured in centimetre
BMI (kg/m^2) | 85 feeding days
  Adolescents BMI (kg/m^2) will be calculated by combining weight and height.

CONTACTS AND LOCATIONS:
Overall Officials: Albert Vandenberg, PhD, Principal Investigator — University of Saskatchewan
Locations (1):
- BRAC Research and Evaluation Division, Dhaka, Bangladesh

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Yunus FM, Jalal C, Das A, Afsana K, Podder R, Vandenberg A, DellaValle DM. Consumption of Iron-Fortified Lentils Is Protective against Declining Iron Status among Adolescent Girls in Bangladesh: Evidence from a Community-Based Double-Blind, Cluster-Randomized Controlled Trial. J Nutr. 2024 May;154(5):1686-1698. doi: 10.1016/j.tjnut.2024.03.005. Epub 2024 Mar 6. PMID 38458577
- [Derived] Yunus FM, Jalal C, Afsana K, Podder R, Vandenberg A, DellaValle DM. Iron-fortified lentils to improve iron (Fe) status among adolescent girls in Bangladesh - study protocol for a double-blind community-based randomized controlled trial. Trials. 2019 May 2;20(1):251. doi: 10.1186/s13063-019-3309-4. PMID 31046819